CLINICAL TRIAL: NCT01981850
Title: A Phase 2, Prospective Study Of PRM-151 In Subjects With Primary Myelofibrosis (PMF), Post-Polycythemia Vera MF (Post-PV MF), Or Post-Essential Thrombocythemia MF (Post-ET MF)
Brief Title: A Phase 2 Study of RO7490677 In Participants With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO42355; PRM-151G-101 (Other: Promedior, Inc.); 2015-001718-80 (EudraCT Number)
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Primary Myelofibrosis; Polycythemia Vera; Post-Essential Thrombocythemia Myelofibrosis
Keywords: fibrosis
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera; Fibrosis | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Stage 1: Cohort 1 Weekly (Experimental): Participants who received no treatment for MF in at least two weeks will be assigned to treatment with single agent RO7490677 at a dose of 10 mg/kg IV on Days 1, 3, 5, 8, 15, and 22 of Cycle 1 and Days 1, 8, 15 and 22 of each subsequent 28 day cycle for six cycles.
  Interventions: Biological: RO7490677
- Stage 1: Cohort 1 Every 4 Weeks (Experimental): Paricipants who received no treatment for MF in at least two weeks will be assigned to treatment with single agent RO7490677 at a dose of 10 mg/kg administered IV on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for six cycles.
  Interventions: Biological: RO7490677
- Stage 1: Cohort 2 Weekly (Experimental): Participants on a stable dose of ruxolitinib for at least 12 weeks, with no improvement in spleen during the last four weeks will be assigned to receive RO7490677 in combination with ruxolitinib at a dose of 10 mg/kg administered IV on Days 1, 3, 5, 8, 15, and 22 of Cycle 1 and Days 1, 8, 15 and 22 of each subsequent 28 day cycle for six cycles.
  Interventions: Biological: RO7490677; Drug: Ruxolitinib
- Stage 1: Cohort 2 Every 4 Weeks (Experimental): Participants on a stable dose of ruxolitinib for at least 12 weeks, with no improvement in spleen during the last four weeks will be assigned to receive RO7490677 in combination with ruxolitinib at a dose of 10 mg/kg administered IV on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for six cycles.
  Interventions: Biological: RO7490677; Drug: Ruxolitinib
- Stage 2: Cohort 1 0.3mg/kg Every 4 Weeks (Experimental): Participants will be treated with single agent RO7490677 at a dose of 0.3 mg/kg IV administered as a 60 minute intravenous infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for nine cycles.
  Interventions: Biological: RO7490677
- Stage 2: Cohort 2 3mg/kg Every 4 Weeks (Experimental): Participants will be treated with single agent RO7490677 at a dose of 3.0 mg/kg IV administered as a 60 minute intravenous infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for nine cycles.
  Interventions: Biological: RO7490677
- Stage 2: Cohort 3 10mg /kg Every 4 Weeks (Experimental): Participants will be treated with single agent RO7490677 at a dose of 10 mg/kg IV administered as a 60 minute intravenous infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for nine cycles.
  Interventions: Biological: RO7490677

INTERVENTIONS:
Biological: RO7490677 — IV infusion
  Other Names: originally called PRM-151, and also known as rhPTX-2
Drug: Ruxolitinib — IV infusion
  Other Names: Jakafi
  Arms: Stage 1: Cohort 2 Every 4 Weeks; Stage 1: Cohort 2 Weekly

SUMMARY:
RO7490677 is an investigational drug that is being developed for possible use in the treatment of myelofibrosis (MF), a disease in which the bone marrow, which is the organ in the body that makes blood cells, is replaced by fibrosis, or excess scar tissue.

The purpose of this study is to gather information on whether RO7490677 has an effect on the MF disease, whether it is safe in patients with MF, and how well it is tolerated.

DETAILED DESCRIPTION:
Stage 1 of this study has completed. Stage 1 was an open-label, Simon two stage, Phase 2 study to determine the efficacy and safety of two different dose schedules of RO7490677 in participants with PMF and post ET/PV MF. There were two treatment cohorts, each assigned to one of two dose schedules receiving either single-agent RO7490677 or RO7490677 in combination with ruxolitinib. Participants were assigned to a weekly or every four week dosing schedule by the investigator.

Stage 2 is a randomized, double-blind Phase 2 study to determine the efficacy and safety of three different doses of RO7490677 in participants with PMF and post ET/PV MF. Participants will be randomized to one of three doses: 0.3 mg/kg, 3.0 mg/kg or 10 mg/kg of RO7490677. This is the second stage of an adaptive design study as defined in FDA Draft Guidance for Industry: Adaptive Design Clinical Trials for Drugs and Biologics, February 2010. Modifications to dose levels, schedule, and regimen have been made in Stage 2 based on data from Stage 1.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥18 years of age at the time of signing the Informed Consent Form (ICF);
2. Participants must voluntarily sign an ICF;
3. Participants must have a pathologically confirmed diagnosis of PMF as per the WHO diagnostic criteria or post ET/PV MF;
4. At least Grade 2 marrow fibrosis according to the WHO Grading of Bone Marrow Fibrosis;
5. Intermediate-1, intermediate -2, or high risk disease according to the IWG -MRT Dynamic International Prognostic Scoring System
6. A bone marrow biopsy must be performed within four weeks prior to Cycle 1 Day 1 treatment to establish the baseline fibrosis score;
7. Participants must not be candidates for ruxolitinib based on EITHER:

   1. Platelet count < 50 x 10e9/L, OR
   2. Hgb < 100 g/L, have received ≥ 2 units PRBC in the 12 weeks prior to study entry, and be intolerant of or had inadequate response to ruxolitinib;
8. Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2. (Appendix F);
9. Life expectancy of at least twelve months;
10. At least four weeks must have elapsed between the last dose of any MF- directed drug treatments for myelofibrosis (including investigational therapies) and study enrollment;
11. Recovery to ≤ Grade 1 or baseline of any toxicities due to prior systemic treatments, excluding alopecia;
12. Women of child bearing potential (WCBP), defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if ≤55 years or 12 months if >55 years, must have a negative serum pregnancy test within four weeks prior to the first dose of study drug and must agree to use adequate methods of birth control throughout the study. Adequate methods of contraception are outlined in the protocol.
13. Ability to adhere to the study visit schedule and all protocol requirements;
14. Must have adequate organ function as demonstrated by the following:

    * ALT (SGPT) and/or AST (SGOT) ≤ 3x upper limit of normal (ULN), or ≤ 4 x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis [EMH] related to MF);
    * Direct bilirubin ≤ 1.5 x ULN; or ≤ 2x ULN (if upon judgment of the treating physician, it is believed to be due to EMH related to MF);
    * Serum creatinine ≤ 2.5 mg/dL x ULN.

Exclusion Criteria:

1. White blood cell count > 25 x 10e9/L or > 10% peripheral blood blasts;
2. Other invasive malignancies within the last 3 years, except non- melanoma skin cancer and localized cured prostate and cervical cancer;
3. History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months;
4. Presence of active serious infection;
5. Any serious, unstable medical or psychiatric condition that would prevent, (as judged by the Investigator) the participant from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study;
6. Known history of human immunodeficiency virus (HIV), or known active hepatitis A, B, or C infection;
7. Organ transplant recipients other than bone marrow transplant;
8. Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (11):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Stanford Cancer Institute, Palo Alto, California
  - Emory Hospital, Atlanta, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mount Sinai Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Providence Health Care, Vancouver, British Columbia
  - The Princess Margaret Cancer Centre, Toronto, Ontario
- Hospital Saint-Louis, Paris, France
- Germany (2):
  - University Medical Center RWTH Aachen, Aachen
  - Johannes Wesling Academic Medical Center, Minden
- Israel (2):
  - Hadassah Medical Centre, Jerusalem
  - Meir Medical Centre, Kfar Saba
- Italy (2):
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Marche Nord Hospital, Pesaro
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Radboud University Medical Center, Nijmegen
- Guy's and St. Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Verstovsek S, Foltz L, Gupta V, Hasserjian R, Manshouri T, Mascarenhas J, Mesa R, Pozdnyakova O, Ritchie E, Veletic I, Gamel K, Hamidi H, Han L, Higgins B, Trunzer K, Uguen M, Wang D, El-Galaly TC, Todorov B, Gotlib J. Safety and efficacy of zinpentraxin alfa as monotherapy or in combination with ruxolitinib in myelofibrosis: stage I of a phase II trial. Haematologica. 2023 Oct 1;108(10):2730-2742. doi: 10.3324/haematol.2022.282411. PMID 37165840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 125 participants were enrolled at sites in 8 different countries.
Pre-assignment Details: One randomized participant in Stage 2 did not receive the study treatment, bringing the total number of treated participants to 124.
Groups:
- Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW): Participants who received no treatment for Myelofibrosis (MF) in at least two weeks were assigned to treatment with single agent PRM-151 at a dose of 10 milligram per kilogram (mg/kg) administered as a 30 minute intravenous (IV) infusion on Days 1, 3, 5, 8, 15, and 22 of Cycle 1 and Days 1, 8, 15 and 22 of each subsequent 28 day cycle for six cycles.
- Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W): Participants who received no treatment for MF in at least two weeks were assigned to treatment with single agent PRM-151 at a dose of 10 mg/kg administered as a 30 minute IV infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for six cycles.
- Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib: Participants on a stable dose of ruxolitinib for at least 12 weeks, with no improvement in spleen during the last four weeks were assigned to receive PRM-151 at a dose of 10 mg/kg administered as a 30 minute IV infusion in combination with daily oral ruxolitinib on Days 1, 3, 5, 8, 15, and 22 of Cycle 1 and Days 1, 8, 15 and 22 of each subsequent 28 day cycle for six cycles.
- Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib: Participants on a stable dose of ruxolitinib for at least 12 weeks, with no improvement in spleen during the last four weeks were assigned to receive PRM-151 at a dose of 10 mg/kg administered as a 30 minute IV infusion in combination with daily oral ruxolitinib on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for six cycles.
- Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W: Participants were treated with single agent PRM-151 at a dose of 0.3 mg/kg administered as a 60 minute IV infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for nine cycles.
- Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W: Participants were treated with single agent PRM-151 at a dose of 3.0 mg/kg administered as a 60 minute IV infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for nine cycles.
- Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W: Participants were treated with single agent PRM-151 at a dose of 10 mg/kg administered as a 60 minute IV infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for nine cycles.
- OLE Stage 1: RO7490677 10 mg/kg IV Q4W: Participants who completed the main phase of treatment moved to the open label extension. They were treated with single agent PRM-151 at a dose of 10 mg/kg administered as an IV infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle.
- OLE Stage 1: RO7490677 10 mg/kg IV Q4W + Ruxolitinib: Participants who completed the main phase of treatment moved to the open label extension. They were treated with PRM-151 at a dose of 10 mg/kg administered as an IV infusion in combination with daily oral ruxolitinib on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle.
- OLE Stage 2: RO7490677 10 mg/kg IV Q4W: Participants who completed 9 cycles of the originally assigned treatment could switch to the open label extension. Participants enrolled received PRM-151 at a dose of 10mg/kg Q4W on days 1, 3, and 5 of first cycle of the open label phase and Day 1 of each subsequent 28 day cycle.
Period: Main Phase Stage 1
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Q4W + Ruxolitinib | OLE Stage 2: RO7490677 10 mg/kg IV Q4W
Started | 8 | 7 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Main Study) | 5 | 5 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Informed Consent Withdrawn | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Various reasons | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Main Phase Stage 2
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Q4W + Ruxolitinib | OLE Stage 2: RO7490677 10 mg/kg IV Q4W
Started | 0 | 0 | 0 | 0 | 33 | 32 | 32 | 0 | 0 | 0
Completed (Main Study) | 0 | 0 | 0 | 0 | 20 | 16 | 15 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 13 | 16 | 17 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 6 | 5 | 7 | 0 | 0 | 0
Not completed — Informed Consent Withdrawn | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Various reasons | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0
Period: Open Label Extension (OLE)
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Q4W + Ruxolitinib | OLE Stage 2: RO7490677 10 mg/kg IV Q4W
Started (Continued in OLE) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 5 | 48
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 5 | 48
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 8
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 19
Not completed — Various reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 9
Not completed — Informed Consent Withdrawn | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Stage 1 & Stage 2 reported separately.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W | Total
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 33 | 32 | 32 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] — Participants in the Main Phase Stage 1 part of the study Population: Main Phase Stage 1 reported separately from Main Phase Stage 2.
  Years
    number analyzed (Participants) | 8 | 7 | 6 | 6 | 0 | 0 | 0 | 27
    (all) | 64.3 (11.4) | 70.7 (6.3) | 66.0 (7.3) | 66.2 (8.6) |  |  |  | 66.7 (8.7)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Participants in the Main Phase Stage 2 part of the study Population: Main Phase Stage 2 reported separately from Main Phase Stage 1.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 33 | 32 | 32 | 97
    (all) |  |  |  |  | 70.6 (7.1) | 70.2 (6.5) | 69.4 (8.9) | 70.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Participants in the Main Phase Stage 1 part of the study Population: Main Phase Stage 1 reported separately from Main Phase Stage 2.
  Participants
    number analyzed (Participants) | 8 | 7 | 6 | 6 | 0 | 0 | 0 | 27
    Female | 5 | 2 | 3 | 5 |  |  |  | 15
    Male | 3 | 5 | 3 | 1 |  |  |  | 12
Sex: Female, Male [Count of Participants; unit: Participants] — Participants in the Main Phase Stage 2 part of the study Population: Main Phase Stage 2 reported separately from Main Phase Stage 1.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 33 | 32 | 32 | 97
    Female |  |  |  |  | 16 | 8 | 11 | 35
    Male |  |  |  |  | 17 | 24 | 21 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants in the Main Phase Stage 1 part of the study Population: Main Phase Stage 1 reported separately from Main Phase Stage 2.
  Participants
    number analyzed (Participants) | 8 | 7 | 6 | 6 | 0 | 0 | 0 | 27
    Hispanic or Latino | 0 | 0 | 1 | 0 |  |  |  | 1
    Not Hispanic or Latino | 8 | 7 | 4 | 6 |  |  |  | 25
    Unknown or Not Reported | 0 | 0 | 1 | 0 |  |  |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants in the Main Phase Stage 1 part of the study Population: Main Phase Stage 1 reported separately from Main Phase Stage 2.
  Participants
    number analyzed (Participants) | 8 | 7 | 6 | 6 | 0 | 0 | 0 | 27
    American Indian or Alaska Native | 0 | 0 | 1 | 0 |  |  |  | 1
    Asian | 0 | 0 | 1 | 0 |  |  |  | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  |  |  | 0
    Black or African American | 1 | 0 | 1 | 0 |  |  |  | 2
    White | 7 | 7 | 3 | 6 |  |  |  | 23
    More than one race | 0 | 0 | 0 | 0 |  |  |  | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants in the Main Phase Stage 2 part of the study Population: Main Phase Stage 2 reported separately from Main Phase Stage 1.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 33 | 32 | 32 | 97
    American Indian or Alaska Native |  |  |  |  | 0 | 0 | 0 | 0
    Asian |  |  |  |  | 0 | 1 | 2 | 3
    Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 | 0 | 0 | 0
    Black or African American |  |  |  |  | 0 | 1 | 0 | 1
    White |  |  |  |  | 33 | 29 | 29 | 91
    More than one race |  |  |  |  | 0 | 0 | 0 | 0
    Unknown or Not Reported |  |  |  |  | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Stage 1 Main Phase: Overall Response Rate (ORR)
Description: ORR was defined as the percent of participants with a response according to the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria. This was defined as those participants who achieved clinical improvement (CI), partial remission (PR), or complete remission (CR) at a post-baseline assessment of treatment response OR had at least stable disease (SD) for three consecutive end-of-cycle response assessments (e.g. Day 1 of the subsequent cycle) in conjunction with improvement in the bone marrow fibrosis score relative to baseline by at least one grade at any time point during the period of stable disease.
Time Frame: Up until and including completion of 6 cycles. Each cycle is 28 days.
Population: The all treated population included all participants who received at least one dose of RO7490667.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
Percentage of Participants | 37.5 [11.11 to 71.08] | 14.3 [0.73 to 52.07] | 33.3 [6.28 to 72.87] | 50.0 [15.32 to 84.68]

2. Primary Outcome: Stage 2 Main Phase: Bone Marrow Response Rate (BMRR)
Description: Response rate was defined as the percent of participants with a reduction in bone marrow fibrosis by at least one grade according to World Health Organization (WHO) criteria from baseline to any time during the study. This was determined by a central adjudication panel of expert hematopathologists, blinded to participant, treatment, and time of biopsy.
Time Frame: Up until and including completion of 9 cycles. Each cycle is 28 days.
Population: The all treated population included all participants randomized and who received at least one administration of the drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 33 | 32 | 32
Percentage of Participants | 30.3 [14.62 to 45.98] | 31.3 [15.19 to 47.31] | 25.0 [10.00 to 40.00]

3. Primary Outcome: Stage 1 Main + Open-Label Extension (OLE): ORR
Description: ORR was defined as the percent of participants with a response according to the IWG-MRT criteria. This was defined as those participants who achieved CI, PR, or CR at a post-baseline assessment of treatment response OR had at least SD for three consecutive end-of-cycle response assessments (e.g. Day 1 of the subsequent cycle) in conjunction with improvement in the bone marrow fibrosis score relative to baseline by at least one grade at any time point during the period of stable disease. Participants who achieved a clinical benefit in the main phase had the opportunity to remain on treatment. The determination of ORR in the main phase is outlined in the arms description below. Participants who didn't achieve a benefit had the opportunity to switch to a different dosing schedule in the OLE phase. The determination of ORR in the OLE phase is outlined in the arms descriptions below.
Time Frame: From cycle 1 day 1 up until cycle 6, day 29 (Main Phase). From cycle 7 day 1 up until study discontinuation or study termination, up to 83 cycles (OLE). Each cycle is 28 days.
Population: The all treated population (main phase + OLE) included all participants who received at least one dose of RO7490667.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- Main Phase Stage 1: RO7490677 10 mg/kg IV QW; OLE: RO7490677 10 mg/kg IV Q4W: Participants were followed through their originally assigned treatment. If a participant achieved a clinical benefit in the main phase, they had the opportunity to remain on treatment. Participants who didn't achieve a clinical benefit had the opportunity to switch to a different dosing schedule in the OLE phase. Participants were not allowed to add ruxolitinib if they had been receiving monotherapy during the main phase.
  Participants who received no treatment for Myelofibrosis (MF) in at least two weeks were assigned to treatment with single agent PRM-151 at a dose of 10 milligram per kilogram (mg/kg) administered as a 30 minute intravenous (IV) infusion on Days 1, 3, 5, 8, 15, and 22 of Cycle 1 and Days 1, 8, 15 and 22 of each subsequent 28 day cycle for 6 cycles (main phase) and on Days 1, 3, and 5 of Cycle 7 and Day 1 of each subsequent 28 day cycle for 83 cycles (OLE).
- Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W; OLE: RO7490677 10 mg/kg IV Q4W: Participants were followed through their originally assigned treatment. If a participant achieved a clinical benefit in the main phase, they had the opportunity to remain on treatment. Participants who didn't achieve a clinical benefit had the opportunity to switch to a different dosing schedule in the OLE phase. Participants were not allowed to add ruxolitinib if they had been receiving monotherapy during the main phase.
  Participants who received no treatment for MF in at least two weeks were assigned to treatment with single agent PRM-151 at a dose of 10 mg/kg administered as a 30 minute IV infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for 6 cycles (main phase) and on Days 1, 3, and 5 of Cycle 7 and Day 1 of each subsequent 28 day cycle for 83 cycles (OLE).
- Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib; OLE: RO7490677 10 mg/kg IV Q4W + Ruxo.: Participants were followed through their originally assigned treatment. If a participant achieved a clinical benefit in the main phase, they had the opportunity to remain on treatment. Participants who didn't achieve a clinical benefit had the opportunity to switch to a different dosing schedule in the OLE phase. Participants could drop ruxolitinib in the OLE, but were not allowed to add ruxolitinib if they had been receiving monotherapy during the main phase.
  Participants on a stable dose of ruxolitinib for at least 12 weeks, with no improvement in spleen during the last four weeks were assigned to receive PRM-151 at a dose of 10 mg/kg administered as a 30 minute IV infusion in combination with daily oral ruxolitinib on Days 1, 3, 5, 8, 15, and 22 of Cycle 1 and Days 1, 8, 15 and 22 of each subsequent 28 day cycle for 6 cycles (main phase) and on Days 1, 3, and 5 of Cycle 7 and Day 1 of each subsequent 28 day cycle for 83 cycles (OLE).
- Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W + Ruxolitinib; OLE: RO7490677 10 mg/kg IV Q4W + Ruxo.: Participants were followed through their originally assigned treatment. If a participant achieved a clinical benefit in the main phase, they had the opportunity to remain on treatment. Participants who didn't achieve a clinical benefit had the opportunity to switch to a different dosing schedule in the OLE phase. Participants could drop ruxolitinib in the OLE, but were not allowed to add ruxolitinib if they had been receiving monotherapy during the main phase.
  Participants on a stable dose of ruxolitinib for at least 12 weeks, with no improvement in spleen during the last four weeks were assigned to receive PRM-151 at a dose of 10 mg/kg administered as a 30 minute IV infusion in combination with daily oral ruxolitinib on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for 6 cycles (main phase) and on Days 1, 3, and 5 of Cycle 7 and Day 1 of each subsequent 28 day cycle for 83 cycles (OLE).
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV QW; OLE: RO7490677 10 mg/kg IV Q4W | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W; OLE: RO7490677 10 mg/kg IV Q4W | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib; OLE: RO7490677 10 mg/kg IV Q4W + Ruxo. | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W + Ruxolitinib; OLE: RO7490677 10 mg/kg IV Q4W + Ruxo.
Number analyzed (Participants) | 8 | 7 | 6 | 6
Percentage of Participants | 50.0 [19.29 to 80.71] | 71.4 [34.13 to 94.66] | 50.0 [15.32 to 84.68] | 66.7 [27.13 to 93.72]

4. Primary Outcome: Stage 2 Main + Open-Label Extension (OLE): BMRR
Description: Defined as the percent of participants with a reduction in bone marrow fibrosis score by at least one grade according to WHO criteria at any time during the study. As determined by a central adjudication panel of expert hematopathologists, blinded to participant, treatment, and time of biopsy. Participants in the main phase had the opportunity to remain on treatment (as outlined in the arms description below). Participants also had the option to switch to the OLE phase after completing 9 cycles of the originally assigned treatment and receive PRM-151 10 mg/kg/Q4W (as outlined in the arms description below).
Time Frame: From cycle 1 day 1 up until cycle 9 day 29 (main phase). From cycle 10 day 1 up until study discontinuation or study termination, up to 51 cycles (OLE). Each cycle is 28 days.
Population: The all treated population (main phase + OLE) included all participants randomized and who received at least one administration of the drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W; OLE: RO7490677 10 mg/kg IV Q4W: Participants were followed through their originally assigned treatment. Participants in the main phase had the opportunity to remain on treatment. Participants also had the option to switch to the OLE phase after completing 9 cycles of the originally assigned treatment as outlined below.
  Participants were treated with single agent PRM-151 at a dose of 0.3 mg/kg administered as a 60 minute IV infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for 9 cycles (main phase) and PRM-151 at a dose of 10 mg/kg on Days 1, 3, and 5 of Cycle 10 and Day 1 of each subsequent 28 day cycle for 51 cycles (OLE).
- Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W; OLE: RO7490677 10 mg/kg IV Q4W: Participants were followed through their originally assigned treatment. Participants in the main phase had the opportunity to remain on treatment. Participants also had the option to switch to the OLE phase after completing 9 cycles of the originally assigned treatment as outlined below.
  Participants were treated with single agent PRM-151 at a dose of 3.0 mg/kg administered as a 60 minute IV infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for 9 cycles (main phase) and PRM-151 at a dose of 10 mg/kg on Days 1, 3, and 5 of Cycle 10 and Day 1 of each subsequent 28 day cycle for 51 cycles (OLE).
- Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W; OLE: RO7490677 10 mg/kg IV Q4W: Participants were followed through their originally assigned treatment. Participants in the main phase had the opportunity to remain on treatment. Participants also had the option to switch to the OLE phase after completing 9 cycles of the originally assigned treatment as outlined below.
  Participants enrolled received PRM-151 at a dose of 10mg/kg Q4W on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for 9 cycles (main phase) and on Days 1, 3, and 5 of Cycle 10 and Day 1 of each subsequent 28 day cycle for 51 cycles (OLE).
Arm/Group | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W; OLE: RO7490677 10 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W; OLE: RO7490677 10 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W; OLE: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 33 | 32 | 32
Percentage of Participants | 30.3 [14.62 to 45.98] | 34.4 [17.92 to 50.83] | 25.0 [10.00 to 40.00]

5. Secondary Outcome: Stage 1 Main Phase: BMRR
Description: Bone marrow response was defined as a reduction in bone marrow fibrosis score by at least one grade from baseline at anytime during the study.
Time Frame: Baseline, Weeks 12 and 24
Population: The all treated population included all participants who received at least one dose of RO7490667.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
Percentage of Participants | 37.5 [3.95 to 71.05] | 14.3 [0.00 to 40.21] | 16.7 [0.00 to 46.49] | 50.0 [9.99 to 90.01]

6. Secondary Outcome: Stage 1 Main Phase: Modified Myeloproliferative Neoplasms Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) Changes
Description: The MPN-SAF TSS total symptom score was the sum of the following 10 items: Filling up quickly when you eat (early satiety), abdominal discomfort, inactivity, Problems with concentration, Worst fatigue, Night sweats, Itching, Bone pain, Fever and Unintentional weight loss last 6 months. The MPN-SAF Total Symptom Score had a possible range of 0 to 100, where a lower score was more favorable. The values reported are the change from baseline scores.
Time Frame: Baseline, beginning of each cycle (Cycle 2 onward). Each cycle is 28 days.
Population: The all treated population included all participants who received at least one dose of RO7490667.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
Score on a scale
  Baseline | 23.1 (19.1) | 16.9 (7.2) | 26.8 (17.1) | 15.3 (10.4)
  Cycle(C)2 Day(D)1: number analyzed (Participants) | 7 | 6 | 6 | 6
  Cycle(C)2 Day(D)1 | -5.3 (12.6) | 5.7 (11.8) | 0.5 (8.8) | -2.0 (5.0)
  C3D1: number analyzed (Participants) | 7 | 7 | 6 | 5
  C3D1 | -9.1 (10.9) | 1.9 (5.3) | -2.7 (14.8) | 4.2 (8.0)
  C4D1: number analyzed (Participants) | 7 | 7 | 6 | 6
  C4D1 | -8.7 (10.7) | 1.0 (8.0) | -7.5 (6.0) | 5.7 (20.9)
  C5D1: number analyzed (Participants) | 5 | 7 | 6 | 6
  C5D1 | -13.2 (13.2) | 2.6 (6.9) | -6.7 (10.6) | 1.5 (13.6)
  C6D1: number analyzed (Participants) | 5 | 5 | 5 | 6
  C6D1 | -12.2 (9.5) | -0.8 (8.3) | -5.4 (6.2) | 4.3 (11.5)
  C6D29: number analyzed (Participants) | 5 | 5 | 4 | 4
  C6D29 | -15.0 (13.7) | -2.2 (5.3) | -5.3 (4.6) | 2.3 (8.8)

7. Secondary Outcome: Stage 2 Main Phase: BMRR
Description: Response rate was defined as the percent of participants with a reduction in bone marrow fibrosis by at least one grade according to World Health Organization (WHO) criteria at any time during the study. This was determined by a central adjudication panel of expert hematopathologists, blinded to participant, treatment, and time of biopsy.
Time Frame: Up until and including completion of 9 cycles. Each cycle is 28 days.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 33 | 32 | 32
Percentage of Participants | 30.3 [14.62 to 45.98] | 31.3 [15.19 to 47.31] | 25.0 [10.0 to 40.00]

8. Secondary Outcome: Stage 2 Main Phase: BMRR - Reduction of Bone Marrow Fibrosis by Visit
Description: Reduction in bone marrow fibrosis score: Reduction of at least one grade from baseline. Bone marrow fibrosis grades according to WHO criteria (as determined by central adjudication).
Time Frame: Day 1 on Cycles 4, 7, 10 and Cycle 9 Day 29. Each cycle is 28 days.
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 33 | 32 | 32
Percentage of Participants
  Cycle(C) 4 Day(D) 1: number analyzed (Participants) | 28 | 25 | 26
  Cycle(C) 4 Day(D) 1 | 10.7 | 24.0 | 19.2
  C7D1: number analyzed (Participants) | 21 | 17 | 19
  C7D1 | 23.8 | 11.8 | 10.5
  C9D29/C10D1: number analyzed (Participants) | 20 | 14 | 15
  C9D29/C10D1 | 30.0 | 21.4 | 13.3

9. Secondary Outcome: Stage 2 Main Phase: Duration of Bone Marrow Improvement
Description: Duration of response was defined as time from first decrease from baseline >= 1 grade to time of return to baseline levels.
Time Frame: From first decrease from baseline of one grade to time of return to baseline levels, up to cycle 9 of 28-day cycles.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 33 | 32 | 32
Weeks | NA [12.0 to NA] — Data was not evaluable as the participants who had bone marrow improvement but did not return to baseline levels at the end of main phase were censored at their last bone marrow assessment in the main phase (the last timepoint in the main phase at which the improvement was still observed). | 12.0 [12.0 to NA] — Data was not evaluable as the participants who had bone marrow improvement but did not return to baseline levels at the end of main phase were censored at their last bone marrow assessment in the main phase (the last timepoint in the main phase at which the improvement was still observed). | 12.1 [11.4 to 13.0]

10. Secondary Outcome: Stage 2 Main Phase: Hemoglobin Improvement
Description: Hemoglobin improvement was measured by the percent of participants with: Red cell transfusion independence (no transfusions for >= 12 consecutive weeks) OR 50% reduction in red blood cell (RBC) transfusions for >= 12 consecutive weeks OR percent of participants with >= 10 g/L and >= 20 g/L increase in hemoglobin for >= 12 consecutive weeks without transfusions (outcome parameter assessed was dependent on baseline hemoglobin/transfusion status).
Time Frame: Up until and including completion of 9 cycles. Each cycle is 28 days.
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 33 | 32 | 32
Percentage of Participants | 15.2 | 15.6 | 6.3

11. Secondary Outcome: Stage 2 Main Phase: Platelet Improvement
Description: Platelet improvement was measured by the percent of participants with: Platelet transfusion independence (no transfusions for >= 12 consecutive weeks) OR 50% reduction in platelets transfusions for >= 12 consecutive weeks OR doubling of baseline platelet count for >= 12 consecutive weeks without platelet transfusions OR platelet count > 50 x 10e9/L for >=12 consecutive weeks without platelet transfusions OR doubling of baseline platelet count for >= 12 consecutive weeks without platelet transfusions OR platelet count > 25 x 10e9/L for >= 12 consecutive weeks without platelet transfusions (outcome parameter assessed is dependent on baseline platelet status).
Time Frame: Up until and including completion of 9 cycles. Each cycle is 28 days.
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 33 | 32 | 32
Percentage of Participants | 27.3 | 34.4 | 37.5

12. Secondary Outcome: Stage 2 Main Phase: Symptom Improvement
Description: Symptom improvement was assessed as the percent of participants with 50% reduction in MPN-SAF TSS from baseline over time. The MPN-SAF TSS total symptom score was the sum of the following 10 items: Filling up quickly when you eat (early satiety), abdominal discomfort, inactivity, Problems with concentration, Worst fatigue, Night sweats, Itching, Bone pain, Fever and Unintentional weight loss last 6 months. The MPN-SAF Total Symptom Score had a possible range of 0 to 100, where a lower score was more favorable.
Time Frame: Up until and including completion of 9 cycles. Each cycle is 28 days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 33 | 32 | 32
Participants
  Cycle(C) 2 Day(D) 1: number analyzed (Participants) | 31 | 31 | 29
  Cycle(C) 2 Day(D) 1 | 5 | 2 | 1
  C3D1: number analyzed (Participants) | 30 | 29 | 28
  C3D1 | 6 | 3 | 2
  C4D1: number analyzed (Participants) | 28 | 29 | 28
  C4D1 | 3 | 4 | 2
  C5D1: number analyzed (Participants) | 24 | 25 | 25
  C5D1 | 5 | 2 | 1
  C6D1: number analyzed (Participants) | 23 | 21 | 25
  C6D1 | 8 | 3 | 3
  C7D1: number analyzed (Participants) | 21 | 18 | 20
  C7D1 | 8 | 5 | 0
  C8D1: number analyzed (Participants) | 20 | 18 | 19
  C8D1 | 5 | 3 | 0
  C9D1: number analyzed (Participants) | 21 | 17 | 17
  C9D1 | 5 | 3 | 1
  C9D29/C10D1: number analyzed (Participants) | 20 | 16 | 13
  C9D29/C10D1 | 5 | 2 | 0

13. Secondary Outcome: Stage 2 Main Phase: Percentage of Participants With Complete Response (CR), Partial Response (PR), Clinical Improvement (CI), Stable Disease (SD), and Progressive Disease (PD) According to IWG-MRT Criteria
Description: Best Overall Response: (CR, PR, CI), SD and PD according to the IWG-MRT Criteria.
Time Frame: Up until and including completion of 9 cycles. Each cycle is 28 days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 33 | 32 | 32
Participants
  CR | 0 | 0 | 0
  PR | 0 | 0 | 0
  CI | 8 | 6 | 2
  SD | 20 | 21 | 26
  PD | 3 | 3 | 4
  Not evaluable | 2 | 2 | 0

14. Other Pre Specified Outcome: Stage 1 Main Phase: Maximum Drug Concentration (Cmax)
Description: Cmax is the maximum observed RO7490677 plasma concentration.
Time Frame: Pre-dose on Cycles(C) 1, 2 and 6, Day(D) 1 and C1 D15. Each cycle is 28 days
Population: The PK population included all participants who received at least one dose of rhPTX-2 and had at least one post-dose total PTX-2 concentration result.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per Milliliter (ug/mL)
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
Micrograms per Milliliter (ug/mL)
  C1D1: number analyzed (Participants) | 7 | 7 | 6 | 6
  C1D1 | 133 (48.4) | 113 (28.1) | 164 (23.9) | 112 (90.4)
  C1D15: number analyzed (Participants) | 7 | 0 | 6 | 0
  C1D15 | 127 (31.9) |  | 126 (27.5) |
  C2D1: number analyzed (Participants) | 7 | 7 | 6 | 6
  C2D1 | 107 (26.9) | 110 (20.9) | 149 (29.1) | 130 (80.2)
  C6D1: number analyzed (Participants) | 5 | 5 | 5 | 6
  C6D1 | 142 (70.0) | 111 (28.0) | 136 (34.1) | 142 (27.4)

15. Other Pre Specified Outcome: Stage 1 Main Phase: Time to Maximum Concentration (Tmax)
Description: Time at which the maximum plasma concentration was observed.
Time Frame: Pre-dose on Cycles(C) 1, 2 and 6, Day(D) 1 and C1 D15. Each cycle is 28 days
Population: as for outcome 14
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
Hour (hr)
  C1D1: number analyzed (Participants) | 7 | 7 | 6 | 6
  C1D1 | 1.12 [1.00 to 2.00] | 1.10 [1.00 to 2.08] | 1.14 [1.00 to 2.25] | 1.13 [1.00 to 5.00]
  C1D15: number analyzed (Participants) | 7 | 0 | 6 | 0
  C1D15 | 1.13 [1.03 to 1.80] |  | 1.65 [1.02 to 2.50] |
  C2D1: number analyzed (Participants) | 7 | 7 | 6 | 6
  C2D1 | 1.10 [1.00 to 3.17] | 1.08 [1.03 to 1.08] | 1.05 [1.00 to 1.32] | 1.44 [1.00 to 9.00]
  C6D1: number analyzed (Participants) | 5 | 5 | 5 | 6
  C6D1 | 2.00 [1.03 to 5.20] | 1.07 [1.00 to 2.03] | 1.17 [1.05 to 5.00] | 1.01 [1.00 to 1.08]

16. Other Pre Specified Outcome: Stage 1 Main Phase: Area Under the Curve up to the Last Measurable Concentration (AUC0-last)
Description: Area under the plasma concentration time curve from time 0 to time of last measurable plasma concentration.
Time Frame: Pre-dose on Cycles(C) 1, 2 and 6, Day(D) 1 and C1 D15. Each cycle is 28 days
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hour/mL
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
ug*hour/mL
  C1D1: number analyzed (Participants) | 7 | 7 | 6 | 6
  C1D1 | 1810 (72.0) | 1690 (26.1) | 2590 (28.7) | 1500 (158.3)
  C1D15: number analyzed (Participants) | 7 | 0 | 6 | 0
  C1D15 | 1460 (142.0) |  | 2590 (187.6) |
  C2D1: number analyzed (Participants) | 7 | 7 | 6 | 6
  C2D1 | 127.3 (904) | 504 (84.7) | 2990 (92.0) | 663 (79.5)
  C6D1: number analyzed (Participants) | 5 | 5 | 5 | 6
  C6D1 | 698 (63.0) | 570 (44.8) | 764 (28.9) | 703 (33.8)

17. Other Pre Specified Outcome: Stage 1 Main Phase: Area Under the Concentration-Time Curve Extrapolated to Infinity (AUC0-inf)
Description: Area under the plasma concentration-time curve from 0-time extrapolated to infinity.
Time Frame: Pre-dose on Cycles(C) 1, 2 and 6, Day(D) 1 and C1 D15. Each cycle is 28 days
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hour/mL
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
ug*hour/mL
  C1D1: number analyzed (Participants) | 3 | 7 | 5 | 3
  C1D1 | 2830 (12.9) | 2050 (29.5) | 2970 (34.9) | 3130 (8.6)
  C1D15: number analyzed (Participants) | 4 | 0 | 4 | 0
  C1D15 | 3450 (2.8) |  | 6060 (23.2) |
  C2D1: number analyzed (Participants) | 3 | 0 | 5 | 0
  C2D1 | 2170 (170.9) |  | 4230 (34.8) |
  C6D1: number analyzed (Participants) | 0 | 0 | 1 | 0
  C6D1 |  |  | 819 (NA) — Geometric Coefficient of Variation could not be calculated from data for a single participant. |

18. Other Pre Specified Outcome: Stage 1 Main Phase: Terminal Elimination Half-Life (T1/2)
Description: Apparent terminal elimination half-life of RO7490677.
Time Frame: Pre-dose on Cycles(C) 1, 2 and 6, Day(D) 1 and C1 D15. Each cycle is 28 days
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
hr
  C1D1: number analyzed (Participants) | 3 | 7 | 5 | 3
  C1D1 | 14.7 (19.2) | 17.2 (23.7) | 16.8 (17.7) | 18.4 (7.9)
  C1D15: number analyzed (Participants) | 4 | 0 | 4 | 0
  C1D15 | 31.2 (45.0) |  | 40.4 (12.6) |
  C2D1: number analyzed (Participants) | 3 | 0 | 5 | 0
  C2D1 | 18.0 (220.6) |  | 30.0 (48.6) |
  C6D1: number analyzed (Participants) | 0 | 0 | 1 | 0
  C6D1 |  |  | 1.95 (NA) — Geometric Coefficient of Variation could not be calculated from data for a single participant. |

19. Other Pre Specified Outcome: Stage 1 Main Phase: Clearance (CL)
Time Frame: Pre-dose on Cycles(C) 1, 2 and 6, Day(D) 1 and C1 D15. Each cycle is 28 days
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hour (L/hr)
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
Litres per hour (L/hr)
  C1D1: number analyzed (Participants) | 3 | 7 | 5 | 3
  C1D1 | 0.258 (9.0) | 0.362 (31.5) | 0.269 (32.9) | 0.233 (33.3)
  C1D15: number analyzed (Participants) | 4 | 0 | 4 | 0
  C1D15 | 0.233 (24.9) |  | 0.147 (35.0) |
  C2D1: number analyzed (Participants) | 3 | 0 | 5 | 0
  C2D1 | 0.382 (229.9) |  | 0.189 (55.5) |
  C6D1: number analyzed (Participants) | 0 | 0 | 1 | 0
  C6D1 |  |  | 1.42 (NA) — Geometric Coefficient of Variation could not be calculated from data for a single participant. |

20. Other Pre Specified Outcome: Stage 1 Main Phase: Volume of Distribution (Vd)
Time Frame: Pre-dose on Cycles(C) 1, 2 and 6, Day(D) 1 and C1 D15. Each cycle is 28 days
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres (L)
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib
Number analyzed (Participants) | 8 | 7 | 6 | 6
Litres (L)
  C1D1: number analyzed (Participants) | 3 | 7 | 5 | 3
  C1D1 | 5.47 (10.9) | 9.00 (28.8) | 6.52 (26.4) | 6.17 (38.9)
  C1D15: number analyzed (Participants) | 4 | 0 | 4 | 0
  C1D15 | 10.5 (62.4) |  | 8.57 (47.6) |
  C2D1: number analyzed (Participants) | 3 | 0 | 5 | 0
  C2D1 | 9.93 (63.0) |  | 8.18 (24.5) |
  C6D1: number analyzed (Participants) | 0 | 0 | 1 | 0
  C6D1 |  |  | 4.01 (NA) — Geometric Coefficient of Variation could not be calculated from data for a single participant. |

21. Other Pre Specified Outcome: Percentage of Participants With Adverse Events (AEs) and Infusion Related Reactions (IRRs)
Description: An AE was defined as any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered investigational product-related. Pre-existing conditions which worsened during the study were also considered as adverse events. IRRs were considerd to be Adverse Events of Special Interest (AESI). Grading was completed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.0.
Time Frame: Baseline up until 6.75 years
Population: The safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Groups:
- OLE Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W): Participants who received no treatment for MF in at least two weeks were assigned to treatment with single agent PRM-151 at a dose of 10 mg/kg administered as a 30 minute IV infusion on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for six cycles.
- OLE Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib: Participants on a stable dose of ruxolitinib for at least 12 weeks, with no improvement in spleen during the last four weeks were assigned to receive PRM-151 at a dose of 10 mg/kg administered as a 30 minute IV infusion in combination with daily oral ruxolitinib on Days 1, 3, and 5 of Cycle 1 and Day 1 of each subsequent 28 day cycle for six cycles.
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | OLE Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib | OLE Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 33 | 32 | 32 | 13 | 5 | 48
Percentage of Participants
  AEs | 100 | 85.7 | 100 | 100 | 100 | 100 | 100 | 92.3 | 100 | 89.6
  IRRs | 0 | 0 | 0 | 16.7 | 3.0 | 3.1 | 6.3 | 7.7 | 20.0 | 2.1

22. Other Pre Specified Outcome: Percentage of Participants With Serious Adverse Events (SAEs) and AEs Leading to Study Drug Discontinuation
Description: An SAE was defined as any AE that occurred at any dose the resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalizations; a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly or birth defect. An AE was defined as any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered investigational product-related. Pre-existing conditions which worsened during the study were also considered as adverse events. Grading was completed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.0.
Time Frame: Baseline up until 6.75 years
Population: The safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | OLE Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib | OLE Stage 2: RO7490677 10 mg/kg IV Q4W
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 33 | 32 | 32 | 13 | 5 | 48
Percentage of Participants
  SAEs | 25.0 | 0 | 0 | 0 | 15.2 | 15.6 | 28.1 | 7.7 | 0 | 22.9
  AEs | 25.0 | 0 | 0 | 0 | 21.2 | 34.4 | 37.5 | 30.8 | 0 | 27.1

ADVERSE EVENTS:
Time Frame: Baseline up until 6.75 years
Description: Treatment-emergent adverse events (TEAEs) were defined as any AE that occurred after the administration of any amount of the study drug, or any event that was present at baseline.
Arm/Group | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Q4W | OLE Stage 1: RO7490677 10 mg/kg IV Q4W + Ruxolitinib | OLE Stage 2: RO7490677 10 mg/kg IV Q4W
All-Cause Mortality (participants affected / at risk) | 2/8 | 0/7 | 1/6 | 0/6 | 7/33 | 6/32 | 9/32 | 0/13 | 0/5 | 7/48
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/7 | 2/6 | 0/6 | 11/33 | 14/32 | 14/32 | 5/13 | 2/5 | 22/48
Other Adverse Events (participants affected / at risk) | 8/8 | 6/7 | 6/6 | 6/6 | 32/33 | 30/32 | 31/32 | 12/13 | 5/5 | 32/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) (N=8) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) (N=7) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib (N=6) | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib (N=6) | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W (N=33) | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W (N=32) | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W (N=32) | OLE Stage 1: RO7490677 10 mg/kg IV Q4W (N=13) | OLE Stage 1: RO7490677 10 mg/kg IV Q4W + Ruxolitinib (N=5) | OLE Stage 2: RO7490677 10 mg/kg IV Q4W (N=48)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Urinary bladder rupture (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every Week (QW) (N=8) | Main Phase Stage 1: RO7490677 10 mg/kg IV Every 4 Weeks (Q4W) (N=7) | Main Phase Stage 1: RO7490677 10 mg/kg IV QW + Ruxolitinib (N=6) | Main Phase Stage 1: RO7490677 10 mg/kg IV Q4W+ Ruxolitinib (N=6) | Main Phase Stage 2: RO7490677 0.3 mg/kg IV Q4W (N=33) | Main Phase Stage 2: RO7490677 3 mg/kg IV Q4W (N=32) | Main Phase Stage 2: RO7490677 10 mg/kg IV Q4W (N=32) | OLE Stage 1: RO7490677 10 mg/kg IV Q4W (N=13) | OLE Stage 1: RO7490677 10 mg/kg IV Q4W + Ruxolitinib (N=5) | OLE Stage 2: RO7490677 10 mg/kg IV Q4W (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (11) | 6 (8) | 3 (6) | 1 (2) | 1 (1) | 6 (12)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (3) | 3 (3) | 0 (0) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 6 (8) | 4 (5) | 1 (1) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 3 (4) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 8 (8) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 7 (7)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 4 (5) | 2 (3) | 3 (5)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 5 (9) | 2 (2) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (3) | 1 (1) | 8 (9) | 8 (10) | 11 (12) | 2 (2) | 0 (0) | 5 (5)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (8) | 3 (4) | 9 (10) | 2 (2) | 0 (0) | 4 (5)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 7 (8) | 3 (3) | 0 (0) | 1 (2) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 3 (3)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 2 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 5 (5)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (7) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (9) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (5) | 4 (6) | 1 (1) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (5) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 2 (2) | 2 (2) | 4 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (9) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 7 (8) | 3 (3) | 2 (3) | 2 (4) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 10 (12) | 7 (8) | 5 (5) | 2 (3) | 3 (4) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (7) | 8 (10) | 7 (8) | 0 (0) | 0 (0) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 5 (7) | 4 (4) | 4 (11) | 0 (0) | 1 (1) | 7 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (4) | 4 (6) | 0 (0) | 0 (0) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 4 (5)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 2 (3) | 0 (0) | 0 (0) | 3 (6)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 8 (8) | 8 (11) | 0 (0) | 0 (0) | 5 (6)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatic nerve neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood product transfusion dependent (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT01981850/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT01981850/SAP_001.pdf